CLINICAL TRIAL: NCT02142400
Title: A Double Blind, Randomised, Placebo-controlled, Multiple Ascending-dose Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of DS 1093a in Healthy Male Subjects
Brief Title: Multiple Ascending Dose Study of DS-1093 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DS1093-A-E102
Record Dates: First submitted 2014-05-14; First posted 2014-05-20 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2015-04

CONDITIONS: Anaemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DS-1093 (Experimental): Group 1 will receive 10mg, group 2 will receive 25mg of DS-1093
  Interventions: Drug: DS-1093
- placebo (Placebo Comparator): placebo to match DS-1093 dosage
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: DS-1093 — DS-1093 in capsules with 2.5mg or 25mg per capsule
  Arms: DS-1093
Drug: placebo — matching placebo capsules to DS-1093 capsules
  Arms: placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled multiple ascending single study. It is hypothesised that at least dose of DS-1093a will be safe and tolerable over a 2-week treatment period and will result in increases in reticulocyte count and haemoglobin concentrations in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects, aged 18-45 years.
* A body mass index (BMI, or Quetelet index) in the range 18.0-30.0
* Willing to use a reliable method of contraception during the trial, and for 4 months afterwards
* Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire trial.
* Willingness to give written consent to participate after reading the information and consent form (ICF), and after having the opportunity to discuss the trial with the Investigator or his delegate.
* Willingness to give written consent to have data entered into The Overvolunteering Prevention System.

Exclusion Criteria:

* Clinically relevant abnormal medical history, physical findings, electrocardiogram (ECG), or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
* Presence of acute or chronic illness or history of chronic illness (particularly hypertension, seizures, kidney disease or liver disease, including known or newly discovered Gilbert's syndrome) sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
* Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of psychotic mental illness.
* Presence or history of malignant disease, other than basal cell carcinoma that was successfully treated at least 5 years ago.
* Any medical history that, in the opinion of the Investigator, is suggestive of a significant bleeding or coagulation risk.
* History of venous or arterial thrombosis or embolic disease.
* History of gastric or duodenal ulcer.
* History of treatment with, or use of, an erythropoiesis stimulating agent (e.g. EPO).
* Blood pressure (BP) and heart rate in supine position at the screening examination outside the ranges 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min.
* Haemoglobin concentration of < 129 g/L, platelets outside the normal reference ranges at the screening examination, or evidence of iron deficiency based on serum iron and ferritin levels.
* Surgery (e.g. stomach bypass) or medical condition that might affect absorption of medicines.
* Presence or history of significant hypersensitive or allergic reaction to any drug, except penicillin.
* Use of a prescription medicine or a strong inducer or inhibitor of cytochrome P450 enzymes, during the 30 days before the first dose of trial medication; use of any other over-the-counter medicine, with the exception of acetaminophen (paracetamol), during the 7 days before the first dose of trial medication.
* Participation in another clinical trial of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical trials during the study and for 3 months after receipt of the final dose of trial medication.
* Positive test for hepatitis B, hepatitis C, HIV 1 & HIV 2.
* Abuse of drugs or alcohol during the 2 years before the first dose of trial medication.
* Evidence of drug or alcohol abuse at screening, or intake of more than 21 units of alcohol weekly.
* Use of tobacco or nicotine-containing products during the 3 months before the first dose of trial medication.
* Loss of more than 400 mL blood, or donation of blood, plasma, platelets, or any other blood components, during the 3 months before the trial, or unwilling to abstain from donating during the study and for 3 months after receipt of the final dose of trial medication.
* Possibility that the volunteer will not cooperate with the requirements of the protocol.
* Objection by General Practitioner (GP) to volunteer entering trial.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
blood concentration of DS-1093 | time of dosing through Day 15
  level of DS-1093 will be determined in participants blood from the time of initial dosing through 15 days after.
number of adverse events including type and severity | date of randomization through Day 98
  number, type and severity of adverse events will be reported during the study from initial randomization through Day 98

SECONDARY OUTCOMES:
levels of EPO | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for EPO (Erythropoietin ) through 42 days after initial dosing
levels of VEGF | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted forVEGF (Vascular Endothelial Growth Factor) through 42 days of dosing.
levels of H25 | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for H25 (Hepcidin-25); through 42 days of dosing.
levels of Reticulocytes | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for hematology markers {RET (Reticulocytes), through 42 days of dosing.
levels of Haemoglobin | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for hematology markers Hb (haemoglobin), through 42 days of dosing.
levels of Haematocrit | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for hematology markers HCT (haematocrit), through 42 days of dosing.
levels of Red Blood Cells | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for hematology marker RBC (red blood cells) through 42 days of dosing.
levels of Serum Iron | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for iron metabolism marker {SI (Serum Iron) through 42 days of dosing.
levels of Transferrin | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for iron metabolism markers T (Transferrin), through 42 days of dosing.
levels of TSAT | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for iron metabolism marker TSAT(Saturated Transferrin) through 42 days of dosing.
levels of Ferrin | time of dosing through 42 days after dosing
  Pharmacodynamic (PD) analyses will be conducted for iron metabolism marker F (Ferritin) through 42 days of dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/